CLINICAL TRIAL: NCT01500681
Title: A Prospective Observational Study of Maintenance Plasma Exchange (PLEX) for Neuromyelitis Optica Spectrum Disorders (MultiPLEX Study)
Brief Title: Maintenance Plasma Exchange for Neuromyelitis Optica
Acronym: MultiPLEX
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Terumo BCT (Industry)
Responsible Party: Principal Investigator, Dean Wingerchuk, Principal Investigator, Mayo Clinic
Other Study IDs: 10-007339; MultiPLEX-2012
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; Recurrent Idiopathic Longitudinally Extensive Transverse Myelitis
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Plasma Exchange

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance PLEX
  Interventions: Procedure: Plasma exchange (PLEX)

INTERVENTIONS:
Procedure: Plasma exchange (PLEX) — Regular maintenance PLEX courses, typically 3 procedures monthly

SUMMARY:
Neuromyelitis optica (NMO) is an inflammatory disease of the central nervous system that is associated with autoantibodies to aquaporin-4. Treatment options for prevention of clinical relapses of NMO include immunosuppressive medications. Plasma exchange (PLEX) is commonly used as a rescue therapy for NMO relapses but ongoing, regular PLEX procedures (maintenance PLEX) is sometimes used to prevent relapses. This observational registry will record feasibility, tolerability, safety, and preliminary efficacy data regarding maintenance PLEX for NMO.

DETAILED DESCRIPTION:
Neuromyelitis optica (NMO) is an inflammatory disease of the central nervous system that is associated with autoantibodies to aquaporin-4. Treatment options for prevention of clinical relapses of NMO include immunosuppressive medications. Plasma exchange (PLEX) is commonly used as a rescue therapy for NMO relapses but ongoing, regular PLEX procedures (maintenance PLEX) is sometimes used to prevent relapses. This observational registry will record feasibility, tolerability, safety, and preliminary efficacy data regarding maintenance PLEX for participants with NMO, NMO spectrum disorders, and recurrent idiopathic longitudinally extensive transverse myelitis.

ELIGIBILITY:
Inclusion Criteria:

* Neuromyelitis optica
* Neuromyelitis optica spectrum disorder
* Recurrent idiopathic longitudinally extensive myelitis
* Age 18 years or greater

Exclusion Criteria:

* Any condition that in the opinion of the investigator could increase a participant's risk by participating in the observational study or confound the outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuromyelitis optica/CNS demyelinating disease specialty clinics
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07-09 (Actual); Study Completion 2015-07-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete planned maintenance PLEX regimen | One year
Number of participants with adverse events | One year
Annualized clinical relapse rate | One year

SECONDARY OUTCOMES:
Median Expanded Disability Status Score (EDSS) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Dean M Wingerchuk, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials